CLINICAL TRIAL: NCT07049991
Title: Para-Prosthetic Valve Leak Closure Observatory - PVLC2
Acronym: FFPP2
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02930-57
Record Dates: First submitted 2025-06-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Para-prosthetic Heart
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical or percutaneous heart valve replacement. — para-prosthetic heart valve leakage after after surgical or percutaneous heart valve replacement

SUMMARY:
Para-prosthetic heart valve leakage is an evolving complication after surgical or percutaneous heart valve replacement. These leaks can lead to heart failure and/or life-threatening hemolysis.

Percutaneous closure of para-prosthetic leaks has developed as an alternative to surgery in high-risk surgical patients. These procedures remain difficult on the technical side with a significant risk of failure and complications but have been improving since the development of dedicated prostheses and the increase in operator experience.

A sharing of experience through the creation of an international expert group has been initiated since 2017 formalised by biannual expert meetings, the elaboration of recommendations in progress and the establishment of an international observatory PVLC1(CCTIRS N°16-62) on 2017-2019.

Beyond the technical aspects and the follow-up of major cardiovascular events collected in PVLC1, the investigators also wonder what impact these procedures have on the quality of life of patients. The investigators suggest that even a partial decrease in para-prosthetic leakage may be associated with an improvement in quality of life by reducing the need for transfusion and/or reducing dyspnea.

A new PVLC2 study is justified to continue the evolutionary follow-up of the technical and clinical results of these procedures, accompanied by the evaluation of the possible benefit on the quality of life of the patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years and older
* Non-opposition of the patient or child's legal representative
* Patient referred for a percutaneous para-prosthetic leakage closure procedure

Exclusion Criteria:

* ≤ 16 years of age
* Refusal of the patient to participate in the observatory or the legal representative if the patient is a minor.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients adressed for a paravalvular leak closure.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the technical and clinical results of the closure of para-prosthetic leaks by assessing the clinical success of the procedure | 2 years
  Clinical success of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Marie Lannelongue Hospital, Le Plessis-Robinson, France